CLINICAL TRIAL: NCT00000677
Title: SCH 39304 as Therapy for Acute Cryptococcal Meningitis in HIV-Infected Patients Followed by Maintenance Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Schering-Plough (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 125; C89-258
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-12

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: Sch 39304; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Drug Evaluation; Antifungal Agents; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Sch 39304

INTERVENTIONS:
Drug: SCH 39304

SUMMARY:
To assess the safety and effectiveness of SCH 39304 as primary treatment of acute cryptococcal meningitis in HIV-infected patients. Safety and effectiveness of maintenance therapy following successful treatment of acute disease are also evaluated.

Cryptococcal meningitis is a significant cause of illness and death in HIV-infected patients. Intravenous amphotericin B is effective for acute disease but relapse occurs in the majority of patients. Maintenance therapy is recommended but must be balanced against the multiple toxicities of the drugs used and the problems associated with the weekly administration of intravenous therapy. Treatments that are equally or more effective and less toxic than traditional methods are needed, especially oral therapy. SCH 39304 is an orally active antifungal drug that in animal studies is active against a wide range of systemic fungal infections including infections due to Cryptococcus. Features of SCH 39304 suggest that it might be of value in the treatment of cryptococcal meningitis.

DETAILED DESCRIPTION:
Cryptococcal meningitis is a significant cause of illness and death in HIV-infected patients. Intravenous amphotericin B is effective for acute disease but relapse occurs in the majority of patients. Maintenance therapy is recommended but must be balanced against the multiple toxicities of the drugs used and the problems associated with the weekly administration of intravenous therapy. Treatments that are equally or more effective and less toxic than traditional methods are needed, especially oral therapy. SCH 39304 is an orally active antifungal drug that in animal studies is active against a wide range of systemic fungal infections including infections due to Cryptococcus. Features of SCH 39304 suggest that it might be of value in the treatment of cryptococcal meningitis.

HIV-infected patients with a diagnosis of acute cryptococcal meningitis, previously untreated or relapsed following a successfully treated acute episode, are enrolled in the study. SCH 39304 is administered orally once daily for 3 days followed by a lower dose once daily for 12 weeks. Patients who respond to primary therapy are randomized to receive SCH 39304 maintenance therapy at a higher dose once weekly or at the lower dose once daily for up to 12 months under this protocol.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Currently approved antiviral therapy.
* Maintenance therapy for cytomegalovirus retinitis or toxoplasmosis.
* Rifampin.
* Isoniazid.
* Dilantin or barbiturates if investigator agrees to rigorously monitor anticonvulsant drug levels.
* Coumarin-type anticoagulants if investigator agrees to rigorously monitor prothrombin time.
* Prophylactic treatment for Pneumocystis carinii pneumonia (PCP).

Concurrent Treatment:

Allowed:

* Local radiotherapy for mucocutaneous Kaposi's sarcoma.

Prior Medication:

Allowed:

* Amphotericin B, up to 1 mg/kg, during the previous 7 days.

Patients must be HIV positive by 2 methodologies and have either primary cryptococcal meningitis with no prior anti-cryptococcal therapy or relapsed disease after prior therapy.

* Prior therapy for cryptococcal meningitis is limited to approved drugs.
* Written informed consent either from patient or patient's parent or legal guardian is required.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of hypersensitivity to imidazole or azole compounds.
* Central nervous system disease.
* Acute opportunistic infection.
* Underlying conditions that in the opinion of the investigator could preclude assessment of response.

Concurrent Medication:

Excluded:

* Systemic antifungal drugs other than study drug.
* Any investigational drug other than treatment IND drugs.
* Oral hypoglycemic agents.
* Oral contraceptives.
* Cytotoxic chemotherapy.

Patients with the following are excluded:

* Unable to take oral medications.
* Concurrent central nervous system disease which in opinion of investigator would interfere with assessment of response.
* Concurrent acute opportunistic infection requiring therapy (patients who develop an acute opportunistic infection after initiation of study medication may remain on study medication).

Prior Medication:

Excluded within 7 days of study entry:

* Amphotericin B, > 1 mg/kg.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: WG Powderly, Study Chair
Locations (28):
- United States (28):
  - Birmingham Veterans Administration Med Ctr, Birmingham, Alabama
  - Dr Robert Larsen, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Med College of Georgia, Augusta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ Hosp, Boston, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Erie County Med Ctr, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Med Ctr, Columbus, Ohio
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Lee BL, Padula AM, Tauber MG, Chambers HF, Sande MA. Oral SCH 39304 as primary, salvage, and maintenance therapy for cryptococcal meningitis in AIDS. J Acquir Immune Defic Syndr (1988). 1992;5(6):600-4. PMID 1588494